CLINICAL TRIAL: NCT02005601
Title: Does Duloxetine Reduce Sub-Acute Pain After Knee Arthroplasty?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012-016
Record Dates: First submitted 2013-12-04; First posted 2013-12-09 (Estimated); Results first posted 2017-08-29 (Actual); Last update posted 2017-08-29 (Actual); Status verified 2017-07

CONDITIONS: Total Knee Arthroplasty
MeSH Terms: interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Duloxetine (Experimental): Patients will receive 60mg of duloxetine per dose. 1 capsule will be taken preoperatively. Starting on postoperative day (POD) 1, patients will take one capsule once a day until end of POD14.
  Interventions: Drug: Duloxetine 60mg
- Control (Placebo Comparator): Patients will receive 0mg of duloxetine
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Patients will receive placebo drug with no active ingredients per dose. 1 capsule will be taken pre-operatively. One capsule once a day until end of POD14.
  Arms: Control
Drug: Duloxetine 60mg — Patients will receive 60mg of duloxetine per dose. 1 capsule will be taken pre-operatively. One capsule once a day until end of POD14.
  Other Names: Cymbalta
  Arms: Duloxetine

SUMMARY:
We are investigating the impact of duloxetine ("Cymbalta"), a serotonin and norepinephrine reuptake inhibitor, on pain after total knee arthroplasty (TKA). Specifically, the investigators will determine whether duloxetine, 60 mg daily for 2 weeks, reduces pain scores 2 weeks after TKA.

ELIGIBILITY:
Inclusion Criteria:

* Patients with osteoarthritis scheduled for primary tricompartmental total knee arthroplasty with a participating surgeon
* Age 25 to 75 years
* Planned use of regional anesthesia
* Ability to follow study protocol
* English speaking (primary outcome obtained via telephone call and secondary outcomes include questionnaires validated in English only)
* Patients planning on being discharged home or to a rehabilitation center that has agreed to participate

Exclusion Criteria:

* Concurrent use of duloxetine or other SNRIs, MAOIs, Tricyclic antidepressants, triptans (sumatriptan, rizatriptan, naratriptan, zolmitriptan, eletriptan, almotriptan, frovatriptan), lithium, buspirone, St. John's Wort
* Hepatic insufficiency
* Renal insufficiency
* Patients younger than 25 years old and older than 75
* Patients intending to receive general anesthesia
* Allergy or intolerance to one of the study medications
* Patients with an ASA of IV
* Chronic gabapentin/pregabalin use (regular use for longer than 3 months)
* Chronic opioid use (taking opioids for longer than 3 months)
* Patients with major prior ipsilateral open knee surgery

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2013-11; Primary Completion 2015-05 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacques T YaDeau, MD, PhD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Duloxetine | Control
Started | 53 | 53
Completed | 53 | 53
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Duloxetine | Control | Total
Number analyzed (Participants) | 53 | 53 | 106
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 67 [61 to 71] | 63 [57 to 67] | 64 [59 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 26 | 54
  Male | 25 | 27 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 50 | 46 | 96
  Unknown or Not Reported | 0 | 4 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 48 | 48 | 96
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 53 | 53 | 106
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m^2] | 31 [27 to 36] | 31 [27 to 35] | 31 [27 to 35]
Knee pain severity with ambulation [Mean (Standard Deviation); unit: Units on a scale] — Knee pain severity assessed on Numeric Pain Rating scale, which range from 0 (no pain) to 10 (worst pain)
  Units on a scale | 5.8 (2.5) | 5.2 (2.6) | 5.5 (2.6)

OUTCOME MEASURES:

1. Primary Outcome: NRS Pain With Ambulation at 2 Weeks
Description: When considering the pain in the knee in which you are having/had surgery, on a scale of 0-10, with 0 being no pain and 10 being pain as bad as you can imagine, how would you describe your level of pain in the last 24 hours during ambulation?
Time Frame: 2 weeks after surgery
Measure: Mean (Standard Deviation); unit: NRS pain score
Arm/Group | Duloxetine | Control
Number analyzed (Participants) | 53 | 53
NRS pain score | 3.5 (2.1) | 3.8 (2.3)

2. Secondary Outcome: Total Daily Opioid Use (mg Oral Morphine Equivalents)
Description: Total daily opioid use (including PO, PCEA, IV, subcutaneous, IV push) in mg oral morphine equivalents on POD 1.
Time Frame: POD 1
Measure: Mean (Standard Deviation); unit: mg oral morphine equivalents
Arm/Group | Duloxetine | Control
Number analyzed (Participants) | 53 | 53
mg oral morphine equivalents | 57.8 (28.4) | 72.7 (34.9)

3. Secondary Outcome: Nausea Severity
Description: Nausea severity measured using Likert scale ranging from 0 (none) to 10 (severe).
Time Frame: POD 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine | Control
Number analyzed (Participants) | 53 | 53
units on a scale | 0.9 (2.2) | 2.3 (3.4)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Duloxetine | Control
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/53
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/53
Other Adverse Events (participants affected / at risk) | 4/53 | 3/53
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine (N=53) | Control (N=53)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Nausea (General disorders) | 2 (2) | 1 (1)
Headache (General disorders) | 0 (0) | 1 (1)
Somnolence (General disorders) | 1 (1) | 0 (0)
SIADH (Endocrine disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes